CLINICAL TRIAL: NCT05389982
Title: Usage of a Mobile Health Platform for Surveillance of Kidney Stone Formers
Brief Title: Mobile Health Platform for Surveillance of Kidney Stone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped early due to lack of recruitment/difficulty meeting recruitment goal.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Director of the Endourology/Stone Division, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00216640
Record Dates: First submitted 2022-05-06; First posted 2022-05-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-03

CONDITIONS: Stone, Kidney
MeSH Terms: conditions — Kidney Calculi | interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (Placebo Comparator)
  Interventions: Other: Standard Care
- standard care + mHealth (GetWell) (Active Comparator)
  Interventions: Other: mHealth (GetWell); Other: Standard Care
- mHealth (GetWell) (Active Comparator)
  Interventions: Other: mHealth (GetWell)

INTERVENTIONS:
Other: mHealth (GetWell) — GetWell Loop utilizes an interactive health care application to allow patients to more actively participate in their care. We plan to work with GetWell to develop a custom build plan for kidney stone formers to achieve key aspects of stone prevention and provide patient education. This care plan will be developed using native capabilities within GetWell Loop.
  Arms: mHealth (GetWell); standard care + mHealth (GetWell)
Other: Standard Care — Office based pathway
  Arms: Standard Care; standard care + mHealth (GetWell)

SUMMARY:
We plan to investigate whether usage of a mobile health platform for surveillance of stone formers by itself or as an adjunct to standard office-appointments will improve patient compliance and adherence to treatment guidelines and ultimately improve patient care, satisfaction, quality of life, and decrease stone recurrence.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* urinary tract stone formers
* meet the AUA guideline indication for metabolic stone evaluation and surveillance
* willing to pursue treatment recommendations of a metabolic workup

Exclusion Criteria:

* patients without mobile phone capability to utilize GetWell Loop,
* physical or cognitive impairment precluding usage of mobile phone or answering of questionnaires
* non-English speaking
* inability to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
change in patient quality of life | 0 to 6 months
  assess this using the validated Wisconsin Stone Quality of Life questionnaire
change in patient quality of life | 0 to 12 months
  assess this using the validated Wisconsin Stone Quality of Life questionnaire
Change in overall stone health scale | 0 to 6 months
  overall stone health scale (Likert 10-point scale with 1 being "very unhappy with current stone health" and 10 being "couldn't be happier about stone health"),
Change in overall stone health scale | 0 to 12 months
  overall stone health scale (Likert 10-point scale with 1 being "very unhappy with current stone health" and 10 being "couldn't be happier about stone health"),

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No